CLINICAL TRIAL: NCT05570643
Title: The Effects of Human Endotoxemia on Functional Capacity of Hematopoietic Stem and Progenitor Cells
Acronym: LPS-BM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL61136.091.17; 2017-3337 (Other: METC Oost Nederland (Ethical Board))
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Sepsis, Endotoxemia, Immunosuppression
Keywords: Sepsis, immunosuppression, systemic inflammation, human endotoxemia, bone marrow stem and progenitor cells, myelopoiesis, monocytes, transciptomics
MeSH Terms: conditions — Sepsis; Endotoxemia | interventions — Lipopolysaccharides; Endotoxins

STUDY DESIGN:
Intervention Model Description: An pilot study to explore the effects of a LPS-challenge on functional capacity and gene expression of human stem and hematopoietic progenitor cells and blood leukocytes. Subjects will be allocated to a LPS group (n=8 healthy volunteers) that will be challenged with endotoxin twice, or to a placebo group (n=4) who will undergo the same study procedures but receive a placebo challenge (NaCl 0.9%).
Masking Description: LPS is a non-investigational product and will only be used as a challenge agent to induce systemic inflammation. Since the effects op LPS-induced systemic inflammation are profound, no masking will be required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LPS group (Experimental): Healthy male volunteers that will receive an intravenous administration of LPS (2ng/kg) twice.
  Interventions: Drug: LPS
- Placebo group (Placebo Comparator): Healthy male volunteers that will receive an intravenous administration of placebo (NaCl 0.9%).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LPS — This is a non-investigational product. LPS is used as challenge agent to achieve a controlled inflammatory state.
  Other Names: Lipopolysaccharide (LPS from Escherichia coli Type O11); Endotoxin
  Arms: LPS group
Drug: Placebo — Injection of NaCl 0.9%.
  Other Names: NaCl
  Arms: Placebo group

SUMMARY:
We will investigate whether human endotoxemia induces changes in human bone marrow cells and their downstream effector cells. To comprehensively investigate underlying mechanisms behind functional and transcriptional changes in these cell types, we will use state-of-the-art systems biology techniques, including single cell transcriptomics (epi)genetics, and metabolomics.

DETAILED DESCRIPTION:
In the present study, we want to further elucidate the mechanisms behind systemic inflammation and endotoxin tolerance in vivo in humans by focusing on functional changes in hematopoietic stem and progenitor cells. Healthy male volunteers will be challenged with endotoxin to evoke a transient systemic inflammatory response. To evaluate the responses over time, blood and bone marrow aspirates will be collected at multiple timepoints. To comprehensively investigate underlying mechanisms behind functional changes, we will use state-of-the-art systems biology techniques, including single cell transcriptomics, epigenetics (e..g. scATACseq), and metabolomic. As such, this study will yield a comprehensive insight into inflammatory signaling in the different compartments of the body and will thereby improve our understanding of systemic inflammation, endotoxin tolerance,and sepsis, possibly revealing new therapeutic targets to improve sepsis outcome.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 and ≤35 yrs
* Male
* Healthy (as confirmed by medical history, examination, ECG, blood sampling)

Exclusion Criteria:

* Use of any medication
* Smoking
* History or signs of atopic syndrome (asthma, rhinitis with medication and/or eczema)
* Known anaphylaxis or hypersensitivity to the non-investigational products or their excipients.
* History or signs of hematological disease (bone marrow dysfunction):
* Thrombocytopenia (<150*10^9/ml) or anemia (hemoglobin < 8.0 mmol/L)
* Abnormalities in leukocyte differential counts
* History, signs or symptoms of cardiovascular disease, in particular:
* Previous spontaneous vagal collapse
* History of atrial or ventricular arrhythmia
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complete left bundle branch block
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as plasma creatinine >120 μmol/l)
* Liver enzyme abnormalities (above 2x the upper limit of normal)
* Medical history of any disease associated with immune deficiency
* CRP > 20 mg/L, WBC > 12x109/L or < 4 x109/L, or clinically significant acute illness, including infections, within 3 weeks before labeling day
* Previous (participation in a study with) LPS administration
* Any vaccination within 3 months prior to labeling day
* Participation in a drug trial or donation of blood 3 months prior to labeling day
* Recent hospital admission or surgery with general anesthesia (<3 months to labeling day)
* Use of recreational drugs within 21 days prior to labeling day
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Change in function and transcriptional pathways | 15 days
  The change in function and transcriptional pathways (gene expression) of hematopoietic progenitor cells and blood leukocytes (using various functional assays and single cell RNAseq) following human endotoxemia.

SECONDARY OUTCOMES:
Change in (Genome-wide) chromatin accessibility | 15 days
  The change in epigenomic profile (chromatin accessibility) of hematopoietic progenitor cells and blood leukocytes (using single cell ATACseq) following human endotoxemia.
Change in cellular metabolism | 15 days
  The change in cellular metabolism of hematopoietic progenitor cells and blood leukocytes (e.g. using Seahorse analyzer, CYTOF) following human endotoxemia.
Change in macrophage activity in the brain | 15 days
  To changes in tissue resident macrophages activity in the brain (assessed using 18F-DPA-714 labeling and PET examinations) following human endotoxemia.
Life-span of blood leukocytes during homeostasis | 8 days
  To assessment of the life-span and transit times of different subsets of leukocytes and their progenitors in the bone marrow of humans at homeostasis (using Deuterium labeling).
Life-span of blood leukocytes during endotoxemia | 8 days
  To determine the life-span and transit times of different subsets of leukocytes and their progenitors in the bone marrow of humans during human endotoxemia (using Deuterium labeling).

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Medicine, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Single cell transcriptional/gene expression data will be shared.
Supporting Information: SAP, Analytic Code
Access Criteria: Bulk RNA-seq and scRNA-seq data for this study can be downloaded from GEO database (https://www.ncbi.nlm.nih.gov/geo/) with the accession number: GSE212093.
  Codes used to perform the data analysis related to this study are available at https://github.com/fkeramati/LPS-SI